# 定坤丹联合复方口服避孕药治疗 PCOS 的有效性及安全性: 一项开放标签、非随机对照临床研究

主要研究单位:广东省妇幼保健院

研究者: 李荔

方案版本号: 1.0

方案版本日期: 2023年1月30日

# 保密声明

本研究方案包含的所有信息的所有权归本项目的研究者所有,仅提供给伦理委员会和相关机构审阅。在未经主要研究者(PI)书面同意,严禁将任何信息告知与本研究无关的第三方。

# 主要研究者方案签字页

主要研究者关于方案的同意书:

我已经认真阅读过本方案,同意方案中所有的内容,并且同意按方案所描述的内容执行。

我明白缺少伦理委员会同意的情况下,研究不得启动;明白需要获得所有参与研究的受试者的知情同意书和相应的记录文件;明白需根据赫尔辛基宣言等伦理原则及临床研究相关法律法规的要求开展研究;明白需完全遵守本单位的相关规定。

研究者签名(手写):

签字日期:

#### 目录

# 研究方案摘要

- 1.研究背景
- 2. 研究目的
- 3. 研究设计
- 4. 随机化与盲法
- 5. 样本量估算
- 6. 受试者招募
- 7. 研究对象
- 8.研究干预
- 9. 研究流程
- 10. 受试者退出研究或终止研究治疗
- 11.评价指标
- 12. 研究物资管理
- 13. 不良事件、严重不良事件、不良反应
- 14. 数据管理
- 15. 统计分析
- 16. 质量控制与质量保障
- 17. 伦理考虑
- 18. 人类遗传资源相关情况
- 19.研究进度

# 研究方案摘要

| 题目 | 定坤丹联合复方口服避孕药治疗 PCOS 的有效性及安全性: 一项<br>开放标签、非随机对照临床研究 |
|---|---|
| 研究目的 | 研究定坤丹应用于多囊卵巢综合征患者的疗效 |
| 研究设计 | 本研究为单中心、非随机对照、开放标签的临床研究 |
| 样本量 | 以血清雄激素评分下降分数作为主要结局指标,利用样本量计算公式。PCOS 患者使用定坤丹联合复方口服避孕药治疗 3 个月经周期,血清雄激素下 0.53nmol/L,单独使用复方口服避孕药治疗 3 个月经周期,血清雄激素下降 0.21nmol/L,在检验水准 α = 0.05 条件下,若取 80%的检验把握度,考虑 20%的脱落率,试验与对照样本量比值为 1,确定研究组和对照组的样本量各为 60 例,共 120 例。 |
| 研究对象 | 诊断标准(参考 2003 年 ESHRE 与 ASRM 联合提出的鹿特丹标准): (1) 高雄激素血症和(或) 其临床表现; (2) 稀发排卵或无排卵; (3) 卵巢多囊性改变: B超检查见一侧或双侧卵巢直径 2-9mm的卵泡≥12 个和(或) 卵巢体积≥10cm3; (4) 符合上述 3 项中任何 2 项者,即可诊断 PCOS。 纳入标准: (1) 诊断为 PCOS 的妇女; (2) 年龄 18-35 岁,处于育龄期; (3) 近 3 个月内未服用任何激素或中药者; 排除标准: |
| | (1)年龄 <18 岁或 >35 岁; |

| - | |
|---|---|
| | (2)近3个月內曾服用激素或中药者; (3)有先天性肾上腺皮质增生、库欣综合征、分泌雄激素的肿瘤者; (4)肝肾功能异常者; (5)既往有血栓性疾病,动脉或静脉血栓栓塞史者;有重大器质性疾病者。 |
| 主要干预措施 | 研究组: 予以口服优思悦(屈螺酮炔雌醇片(II))治疗,于月经期第1天起按照包装指示服用优思悦(拜耳医药保健有限公司;国药准字: H20140972;规格: 屈螺酮 3mg 和炔雌醇(β-环糊精包合物)0.02mg),每日约在同一时间段内服用,连续服用 28 天,停药后月经来潮,在月经第一天开始下一个用药周期,或予以口服达英-35(决雌醇环丙孕酮片)治疗,于月经期第1天起按照包装指示服用达英-35(拜耳医药保健有限公司;国药准字:注册证号J20100003;规格: 2mg 醋酸环丙孕酮和 0.035mg 炔雌醇),每日约在同一时间段内服用,连续服用 21 天,停药 7 天开始下一个用药周期;在服用复方口服避孕药的同时加定坤丹浓缩水蜜丸(山西国普远有限公司,国药准字: Z20059003,规格: 7g/瓶),每次 3.5g,每日两次。 对照组: 予以口服优思悦(屈螺酮炔雌醇片(II))或予以口服达英-35(决雌醇环丙孕酮片)治疗。 |
| 随访 | 受试者来院复诊,由研究者进行随访追踪;或由研究者通过电话或 微信对受试者进行随访追踪。 |
| 评价指标 | 主要终点指标:血清性激素六项、游离睾酮、雄烯二酮、性激素结合球蛋白;空腹血糖、空腹胰岛素、HOMA-IR; AMH; 同型半胱氨酸; 卵泡发育情况(排卵时卵泡直径); 子宫内膜厚度(卵泡达最大直径时)。 |

| | 次要终点指标:停药后3个月内的周期排卵率、妊娠率、流产率; 肝肾功能及用药后出现不良反应情况。 |
|---|---|
| 统计学方法 | 采用 SPSS 25.0 软件进行统计学分析。计量资料满足正态分布时以 x ±s 表示,组间比较采用两独立样本 t 检验,组内治疗前和治疗 3 个 月经周期后两组比较采用配对 t 检验,血清雄激素比较采用重复测量方差分析;不满足正态分布时以 M (P25, P75)表示,采用非参数秩和检验。计数资料以率或构成比表示,组间比较采用 x 2 检验。P<0.05 为差异有统计学意义。 |
| 研究时间 | 预计首例受试者入组时间: 2023 年 1 月<br>预计最后 1 例受试者入组时间: 2023 年 12 月<br>预计研究结束时间: 2023 年 12 月 |

#### 1、研究背景:

多囊卵巢综合征 (polycystic ovary syndrome, PCOS) 是育龄期女性最常见的妇科内分泌紊乱疾病,患病率约为 5%~10%。PCOS 的危害包括对 PCOS 患者本身以及子代两个方面。首先,PCOS 不但会影响妇女的生殖功能,且增加妇女的代谢障碍(例如:腹型肥胖、血脂异常、血糖稳态受损)和罹患心血管疾病的风险。其次,PCOS 妇女的妊娠相关并发症(例如妊娠糖尿病、高血压疾病、早产等)风险明显增加。再者,有研究发现 PCOS 患者的子代有更高的早产率、围产儿死亡率、和产后住院率,而且其子代更易罹患哮喘、先天畸形、代谢紊乱、心血管疾病。屈螺酮诀雌醇片(II)和诀雌醇环丙孕酮片是西医常用的复方口服避孕药,临床上常用于治疗多囊卵巢综合征,其在帮助建立规律的月经周期和降低雄激素方面有确切的疗效,但停药后病情容易反复发作,且长期服用此药物对患者的肝肾功能及心血管功能不利,故临床上需要去探寻一种更长期、更安全的治疗方案。

定坤丹由当归、香附、柴胡、川芎等 30 味中药材组成,具有滋补气血、调节月经、提高卵巢功能、疏肝止痛的作用,常用于治疗气血两虚、气滞血瘀所致的妇科疾病,如痛经、月经不调、不孕症、更年期综合征和产后诸虚。

如今国内已有一些研究表明,定坤丹联合促排卵药物对 PCOS 不孕的临床效果优于单一使用促排卵药物,使血清 FSH、E2、LH 及 T 等性激素水平降低,并且研究组患者的成熟卵泡直径和子宫内膜厚度都优于对照组,且研究组的妊娠率高于对照组。但国内关于定坤丹治疗 PCOS 的研究仍然很少,且尚无大样本量的 PCOS 患者口服复方口服避孕药联合定坤丹与单独使用复方口服避孕药的临床研究。本研究旨在观察定坤丹对 PCOS 的疗效,为日后中西医联合用药治疗 PCOS 提供更确切的依据。

#### 2、研究目的

(1) 主要目的:研究定坤丹对多囊卵巢综合征患者的疗效,主要对比定坤 丹联合复方口服避孕药与单独使用复方口服避孕药对于降低雄激素的效果、对 患者卵巢功能的影响及对代谢的影响,纳入指标包括血清性激素六项、游离睾酮、雄烯二酮、性激素结合球蛋白; AMH、卵泡发育情况(排卵时卵泡直径); 子宫内膜厚度(卵泡达最大直径时)、空腹血糖、空腹胰岛素、HOMA-IR; 同型半胱氨酸。

(2)次要目的:研究定坤丹对多囊卵巢综合征患者妊娠的影响以及其安全性,纳入指标包括周期排卵率、妊娠率、流产率以及肝肾功能及用药后出现不良反应情况

## 3、研究设计

本研究为单中心、非随机对照、开放标签的临床研究。

# 4、随机化与盲法

无

# 5、样本量估算

以血清雄激素评分下降分数作为主要结局指标,利用样本量计算公式。 PCOS 患者使用定坤丹联合复方口服避孕药治疗 3 个月经周期, 血清雄激素下降 0.53nmol/L;单独使用复方口服避孕药治疗 3 个月经周期,血清雄激素下降 0.21nmol/L,在检验水准  $\alpha=0.05$  条件下,若取 80%的检验把握度,考虑 20%的脱落率,研究与对照样本量比值为 1,确定研究组和对照组的样本量各为 60 例,共 120 例。

#### 6、受试者招募

由研究者在广东省妇幼保健院妇科及妇女保健科招募确诊为 PCOS 育龄期 妇女。

#### 7、研究对象

# 7.1 诊断标准

(1) 高雄激素血症和(或) 其临床表现;

- (2) 稀发排卵或无排卵;
- (3) 卵巢多囊性改变: B 超检查见一侧或双侧卵巢直径 2-9mm 的卵泡≥ 12 个和(或) 卵巢体积≥10cm³;
  - (4) 符合上述 3 项中任何 2 项者,即可诊断 PCOS。

# 7.2 入选标准

- (1) 诊断为 PCOS 的妇女:
- (2) 年龄 18-35 岁, 处于育龄期;
- (3) 近3个月内未服用任何激素或中药者;

#### 7.3 排除标准

- (1) 年龄 < 18 岁或 > 35 岁;
- (2) 近3个月内曾服用激素或中药者;
- (3) 有先天性肾上腺皮质增生、库欣综合征、分泌雄激素的肿瘤者:
- (4) 肝肾功能异常者;
- (5) 既往有血栓性疾病,动脉或静脉血栓栓塞史者,有重大器质性疾病者。

#### 8、研究干预

研究组: 予以口服优思悦(屈螺酮炔雌醇片(II))治疗,于月经期第1天 起按照包装指示服用优思悦(拜耳医药保健有限公司: 国药准字:

H20140972; 规格: 屈螺酮 3mg 和炔雌醇(β-环糊精包合物)0.02mg),每日约在同一时间段内服用,连续服用28天,停药后月经来潮,在月经第一天开始下一个用药周期,在服用复方口服避孕药的同时加定坤丹浓缩水蜜丸(山西国誉远有限公司,国药准字: Z20059003,规格:7g/瓶),每次3.5g,每日两次。

对照组: 予以口服优思悦(屈螺酮炔雌醇片(II))治疗。

两组均连续服药3个月为一个疗程

# 9、研究流程

# (1) 筛选阶段:

2023-1-1 至 2023-12-31 筛选入组患者: 筛选临床确诊为 PCOS 的育龄期且有生育意愿的女性,治疗前 3 个月未使用过相关治疗药,排除有先天性肾上腺皮质增生、库欣综合征、分泌雄激素的肿瘤者,或肝肾功能异者,或既往有血栓性疾病者,或动脉或静脉血栓栓塞史者,或有重大器质性疾病者。

## (2) 随机阶段:

将入组患者分为研究组/对照组,研究组给予复方口服避孕药+定坤丹。对 照组给予复方口服避孕药。

# (3) 治疗阶段:

研究组: 予以口服优思悦(屈螺酮炔雌醇片(II))治疗,于月经期第1天 起按照包装指示服用优思悦(拜耳医药保健有限公司;国药准字:

H20140972; 规格: 屈螺酮 3mg 和炔雌醇(β-环糊精包合物)0.02mg),每日约在同一时间段内服用,连续服用28天,停药后月经来潮,在月经第一天开始下一个用药周期,在服用复方口服避孕药的同时加定坤丹浓缩水蜜丸(山西国誉远有限公司,国药准字: Z20059003,规格:7g/瓶),每次3.5g,每日两次。

对照组: 予以口服优思悦(屈螺酮炔雌醇片(II))治疗。

两组均连续服药3个月为一个疗程

#### (4) 随访阶段:

干预治疗后评估1次,干预治疗3月后再评估1次。





主要结局指标:血清雄激素、雄烯二酮、游离睾酮、性激素结合球蛋白;空腹血糖、空腹胰岛素、HOMA-IR; AMH; 同型半胱氨酸;卵泡发育情况(排卵时卵泡直径);子宫内膜厚度(卵泡达最大直径时)

次要结局指标:周期排卵率、妊娠率、流产率

安全性指标: 肝肾功能及用药后出现不良反应情况。

随访患者3个月内的周期排卵率、妊娠率、流产率。

# 10、受试者退出研究或终止研究治疗

# 10.1 退出研究标准

- (1) 受试者撤回知情同意, 拒绝进一步随访;
- (2) 受试者失访;
- (3) 受试者死亡;

# 10.2 终止研究治疗的标准

- (1) 受试者撤回知情同意,拒绝继续接受研究药物治疗;
- (2) 经研究者判断,受试者临床症状恶化/体力状况下降;

- (3) 经研究者判断,受试者已经达到研究终点;
- (4) 毒性不可耐受,包括出现任何临床 AE、实验室检查异常或其他医疗状况:
  - (5) 研究者认为其他有必要终止研究药物治疗的情况;
  - (6) 研究发起人终止研究。

## 11、评价指标

- (1) 主要观察指标: 血清性激素六项、游离睾酮、雄烯二酮、性激素结合球蛋白; 空腹血糖、空腹胰岛素、HOMA-IR; AMH; 同型半胱氨酸; 卵泡发育情况(排卵时卵泡直径); 子宫内膜厚度(卵泡达最大直径时);
  - (2) 次要观察指标: 停药后3个月内的周期排卵率、妊娠率、流产率。
  - (3) 安全性指标: 肝肾功能及用药后出现不良反应情况。
- 12、研究物资管理(如: 药物、器械、试剂盒等:)

无

# 13、不良事件、严重不良事件、不良反应

服用优思悦可能出现胃肠道不适,如恶心、呕吐、食欲下降等;或(和)子宫不规则出血;或(和)乳房胀痛。研究组和对照组服药后若出现严重不良反应均停止用药,停药后观察不良反应是否消失或减轻,保证受试者得到及时、适当的临床诊治。

#### 14、数据管理

- (1) 2023-1-1 至 2023-12-31,由广东省妇幼保健院负责收集相关数据并记录:
- (2) 2024-1-1 至 2024-1-31,对数据进行整理,对有质疑数据和修改临床试验中所有观察到的结果和异常发现,及时加以认真核实、记录,保证数据的可靠性。

(3) 2024-2-1 至 2024-5-1, 对数据进行统计分析, 得出结论并书写报告。

采用 SPSS 25.0 软件进行统计学分析。计量资料满足正态分布时以 x±s 表示,组间比较采用两独立样本 t 检验,组内治疗前和治疗 3 个月经周期后两组比较采用配对 t 检验,血清雄激素比较采用重复测量方差分析;不满足正态分布时以 M (P25, P75)表示,采用非参数秩和检验。计数资料以率或构成比表示,组间比较采用 x 2 检验。P<0.05 为差异有统计学意义。

## 15、统计学分析

采用 SPSS 25.0 软件进行统计学分析。计量资料满足正态分布时以 x±s 表示,组间比较采用两独立样本 t 检验,组内治疗前和治疗 3 个月经周期后两组比较采用配对 t 检验,血清雄激素比较采用重复测量方差分析;不满足正态分布时以 M (P25, P75)表示,采用非参数秩和检验。计数资料以率或构成比表示,组间比较采用 x 2 检验。P<0.05 为差异有统计学意义。

# 16、质量控制与质量保障

#### 16.1 标准操作规程制定

该研究开展前需进行项目中心启动会,统一多囊卵巢综合征的诊断标准,统一患者纳入、排除标准,统一用药疗程与用药后各项结局指标检测时间。

#### 16.2 参研人员培训和授权分工

研究开展前开展前需对研究者进行统一标准化培训,培训内容包括用药方法、观察指标、不良反应/事件的判断和处理、严重不良事件及不良反应的上报等。

#### 16.3 文档\物资\标本管理

研究者必须充分、准确地记录研究过程,以使研究数据可被核实。这些文件可分成两类,一是研究文件,二是患者的原始数据。研究文件包括方案及其修订、知情同意书样本、研究人员简历和授权表、其它必备的文件和往来信函。

患者的原始文件包括患者住院/门诊的记录,医生和护士的医嘱、预约随访 日期、原始化验报告单、超声检查、签署的知情同意书、患者筛选表等。

# 16.4 受试者依从性管理

认真合理筛选受试者,应诊断准确,对受试者进行全面了解、依从性预评估、仔细筛选,选择依从性佳的受试者,有选择地纳入受试者。充分知情同意过程:签署知情同意书前要求研究者以通俗易懂的语言向受试者及家属进行充分的细的知情说明,让受试者对该试验药物和治疗过程全面了解,对受试者的相关问题进行认真解答,尊重受试者在充分知情的情况下做出的选择,增强受试者完成试验的信心,提高受试者依从性。创造良好的医护患关系,及时妥善处理药物不良事件(AE)与严重不良事件(SAE)。

## 17、伦理考虑

本临床研究遵循赫尔辛基宣言和中国有关临床试验法规进行,在获得伦理委员会批准后方可实施。临床研究期间涉及的临床研究方案、知情同书等资料的修改,需经伦理委员会审批同意后方可执行。研究者需保护受试者的权益和安全,保护受试者的隐私。

# 18、人类遗传资源相关情况

人类遗传资源材料是指含有人体基因组、基因等遗传物质的器官、组织、细胞等遗传材料。人类遗传资源信息是指利用人类遗传资源材料产生的数据等信息资料。

## 19、研究进度

- (1) 2023-1-1 至 2023-12-31,由广东省妇幼保健院负责收集相关数据并记录;
- (2) 2024-1-1 至 2024-1-31,对数据进行整理,对有质疑数据和修改临床试验中所有观察到的结果和异常发现,及时加以认真核实、记录,保证数据的可靠性。

(3) 2024-2-1 至 2024-5-1, 对数据进行统计分析, 得出结论并书写报告。

# 20、参考文献

- [1]宋颖,李蓉.多囊卵巢综合征中国诊疗指南解读[J].实用妇产科杂志,2018,34(10):737-741.
- [2] ESPCW Group. Revised 2003 consensus on diagnostic criteria and longterm health risks related to polycystic ovary syndrome (PCOS) [J]. Fertility Sterility, 2004, 81 (1):41-47.
- [3]Pinola, Pekka et al. "Normo- and Hyperandrogenic Women with Polycystic Ovary Syndrome Exhibit an Adverse Metabolic Profile through Life." Fertility and sterility 107.3 (2016): 788 795.e2.
- [4]Shorakae S, Teede H, de Courten B, Lambert G, Boyle J, Moran LJ. The Emerging Role of Chronic Low-Grade Inflammation in the Pathophysiology of Polycystic Ovary Syndrome. Semin Reprod Med. 2015 Jul;33(4):257-69.
- [5]多囊卵巢综合征相关不孕治疗及生育保护共识[J].生殖医学杂志,2020,29(07):843-851.
- [6]胥杜娟,王安,李琳,向延芳.定坤丹联合来曲唑治疗多囊卵巢综合征不孕的临床效果观察[J]. 中国妇幼保健,2022,37(24):4638-4641.

[7]张玥,孙丹丹,朱加娟,沈炳秋.定坤丹联合西药治疗 PCOS 不孕症的疗效及卵巢储备功能的影响[J/OL].中药材,2022(06):1509-1512[2022-12-28].

[8]徐思敏,胡瑞学,戴泽琦,李慧敏,孙伟伟,廖星.定坤丹治疗女性不孕的疗效评价: 一项基于随机对照试验的系统综述[J].中国实验方剂学杂志,2022,28(08):239-247.